CLINICAL TRIAL: NCT02599909
Title: Gut Microbiota in Patients With HCC
Brief Title: Gut Microbiota in People With Hepatocellular Carcinoma (HCC)
Status: Withdrawn | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916012; 16-C-N012
Record Dates: First submitted 2015-11-06; First posted 2015-11-09 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09-14

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer; Liver Cell Caricinoma; Liver Neoplasm
Keywords: Tumor Microenvironment; 100 Trillion Microbial Cells; Liver Tumors; Intestinal Microbiota; Immune Regulation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1/ Cohort 1: Subjects with hepatocellular carcinoma

SUMMARY:
Background:

There are about 100 trillion microbial cells in a person s gut. This is called the human gut microbiota. When this is disrupted, it can lead to many diseases. Studies show that the gut microbiota in people with cancer is different than that found in healthy people. Researchers want to study links between the gut microbiota and the immune system in people with a liver disease called hepatocellular carcinoma (HCC).

Objective:

To study links between gut microbiota and the immune system in people with HCC.

Eligibility:

People at least 18 years old with HCC. They must be scheduled to have tumors removed by surgery.

Design:

* People having surgery for primary liver tumors at the Mount Sinai Medical Center will be screened for this study.
* At the initial visit, blood, rectal swabs, urine, and stool will be collected. Participants will answer questions about their medical condition.
* Before surgery, blood, rectal swabs, urine, and stool will be collected. This will be done at a routine visit.
* When they have surgery, a piece of liver tissue with the tumor will be collected. This will be sent to the National Cancer Institute for tests.
* After surgery, blood, rectal swabs, urine, and stool will be collected 3 times. This will be done at routine visits.

DETAILED DESCRIPTION:
Background:

The human gut microbiota consists of approximately 100 trillion microbial cells whose disruption leads to many diseases including inflammatory bowel disease and colorectal cancer to name a few. Recent studies have shown that cancer patients have an altered gut microbiota when compared to healthy controls. Intestinal microbiota has been proposed to contribute to the start and progression of a number of liver diseases, such as alcoholic liver disease (ALD), nonalcoholic steatohepatitis (NASH), liver cirrhosis, hepatic encephalopathy (HE), and hepatocellular carcinoma (HCC). We plan to investigate the relationship between the gut microbiota and the immune system in patients with HCC. In recent years, immune regulation at the level of the tumor microenvironment has become very important in different types of cancer.

Objectives:

To collect blood/stool/urine/tumor samples and rectal swabs from HCC patients undergoing resection of primary liver tumors at the Mount Sinai Medical Center and to perform an analysis of the interaction of tumors, immune responses and the gut microbiome.

Eligibility:

* Patients 18 years of age and older
* Patients undergoing liver resection for primary liver cancer
* Patients must be willing to provide informed consent

Design

* Blood, stool, rectal swabs, urine and/or tumor samples may be collected from consenting subjects seen at Mount Sinai Medical Center at the initial visit and/or at follow-up visits.
* Tumor samples will only be obtained from patients undergoing surgery.
* Patients will be asked to answer a questionnaire.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients 18 years of age and older
  2. Patients undergoing a planned resection of hepatocellular carcinoma
  3. Patients must be willing to provide informed consent

EXCLUSION CRITERIA:

Patients with known inflammatory bowel disease or receiving systemic anti-inflammatory treatment.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-06; Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
To collect blood/urine/tumor samples, stool, and rectal swabs from HCC patients undergoing resection of primary liver tumors at the Mount Sinai Medical Center and to perform an analysis of the interaction of tumors, immune responses and the gut ... | 1 year
  Analysis of the interaction of tumors, immune responses and the gut microbiome

SECONDARY OUTCOMES:
Novel mechanisms how tumors may affect immune responses and gut microbiota | 1 year
Correlation between microbiome and patients' clinical outcome | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Goel A, Gupta M, Aggarwal R. Gut microbiota and liver disease. J Gastroenterol Hepatol. 2014 Jun;29(6):1139-48. doi: 10.1111/jgh.12556. PMID 24547986
- [Background] Qin N, Yang F, Li A, Prifti E, Chen Y, Shao L, Guo J, Le Chatelier E, Yao J, Wu L, Zhou J, Ni S, Liu L, Pons N, Batto JM, Kennedy SP, Leonard P, Yuan C, Ding W, Chen Y, Hu X, Zheng B, Qian G, Xu W, Ehrlich SD, Zheng S, Li L. Alterations of the human gut microbiome in liver cirrhosis. Nature. 2014 Sep 4;513(7516):59-64. doi: 10.1038/nature13568. Epub 2014 Jul 23. PMID 25079328
- [Background] De la Fuente M, Franchi L, Araya D, Diaz-Jimenez D, Olivares M, Alvarez-Lobos M, Golenbock D, Gonzalez MJ, Lopez-Kostner F, Quera R, Nunez G, Vidal R, Hermoso MA. Escherichia coli isolates from inflammatory bowel diseases patients survive in macrophages and activate NLRP3 inflammasome. Int J Med Microbiol. 2014 May;304(3-4):384-92. doi: 10.1016/j.ijmm.2014.01.002. Epub 2014 Feb 6. PMID 24581881